CLINICAL TRIAL: NCT05443334
Title: A Multi-centre, Prospective, Non-interventional Single-arm Study Investigating Clinical Parameters Associated With the Use of Once-daily Oral Semaglutide in a Real-world Adult Population With Type 2 Diabetes in Spain
Brief Title: A Research Study Looking at How Oral Semaglutide Works in People With Type 2 Diabetes in Spain, as Part of Local Clinical Practice
Acronym: PIONEER REAL
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9924-4547; U1111-1240-4149 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with type 2 diabetes: Participants with type 2 diabetes and naive to injectable glucose-lowering treatment.
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — Participants will be treated with commercially available oral semaglutide according to local label and to routine clinical practice at the discretion of the treating physician. The decision to initiate treatment with commercially available oral semaglutide has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician based on local label before and independently from the decision to include the participant in this study.

SUMMARY:
The purpose of the study is to collect information on participant's blood sugar levels, body weight, how satisfied participant is with the treatment, and how participant takes his/her diabetes medicines. Participant will get Rybelsus® as prescribed by study doctor. The study will last for about 8-10 months. Participants will be asked to complete a questionnaire about how they take their Rybelsus® tablets. Participants will complete this questionnaire during their normally scheduled visit with the study doctor.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol)
* Diagnosed with type 2 diabetes mellitus
* The decision to initiate treatment with commercially available oral semaglutide has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician based on local label before and independently from the decision to include the patient in this study
* Male or female, age above or equal to 18 years at the time of signing informed consent
* Available HbA1c value less than or equal to 90 days prior to the 'Informed Consent and Treatment Initiation visit' (V1) or HbA1c measurement taken in relation with the 'Informed Consent and Treatment Initiation visit' (V1) if in line with local clinical practice
* Treatment naive to injectable glucose-lowering drug(s). An exception is short-term insulin treatment for acute illness for a total of less than 14 days

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study
* Treatment with any investigational drug within 30 days prior to enrolment into the study
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with type 2 diabetes and naive to injectable glucose-lowering treatment.
Sampling Method: Non-Probability Sample
Enrollment: 465 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2024-07-04 (Actual); Study Completion 2024-07-04 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | From baseline (week 0) to End of Study visit (V3) (week 34-44)
  Measured in percentage (%)-points

SECONDARY OUTCOMES:
Relative change in body weight | From baseline (week 0) to End of Study visit (V3) (week 34-44)
  Measured in percentage (%)
Absolute change in body weight | From baseline (week 0) to End of Study visit (V3) (week 34-44)
  Measured in Kilogram (Kg)
HbA1c < 7% | End of Study visit (V3) (week 34- 44)
  Measured as Yes or No
HbA1c reduction >=1%-points and body weight reduction of >=5% | From baseline (week 0) to End of Study visit (V3) (week 34-44)
  Measured as Yes or No
HbA1c reduction >=1%-points and body weight reduction of >=3% | From baseline (week 0) to End of Study visit (V3) (week 34-44)
  Measured as Yes or No
DTSQc, relative treatment satisfaction | End of Study visit (V3) (week 34- 44)
  Measured in Total score
DTSQs, change in absolute treatment satisfaction | From baseline (week 0) to End of Study visit (V3) (week 34-44)
  Measured in Total score

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (2):
- Spain (2):
  - Master Centre for Spain, Barcelona
  - Master Centre for Spain, Madrid

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Delgado Alvarez E, Morales Portillo C, Abreu Padin C, Aliaga Verdugo A, Piera Carbonell A, Cadenas Gonzalez A, Amor Valero J, Gonzalez Lopez V, Rasmussen CL, Scheuer SH, Bellido Guerrero D. PIONEER REAL Spain: A multicentre, prospective, real-world study of oral semaglutide use in adults with type 2 diabetes. Diabetes Obes Metab. 2025 Sep;27(9):4812-4824. doi: 10.1111/dom.16523. Epub 2025 Jun 24. PMID 40555703